CLINICAL TRIAL: NCT02309970
Title: Perfusion Computer Tomography: Imaging and Clinical Validation Following Reperfusion Therapy in Acute Ischaemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Guy Raphaeli, Dr. Guy Raphaeli, Rabin Medical Center
Other Study IDs: GR 05 - 14
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; apixaban; Rivaroxaban; Dabigatran; Clopidogrel; Warfarin; Acenocoumarol; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Conservative: patient will get treatment with Antiplatelets or Anticoagulant depending on their clinical status/etiology
  Interventions: Drug: acetylsalicylic acid, clopidogrel bisulfate and/or warfarin, Apixaban, Rivaroxaban, Dabigatran
- IV tPA: patient will receive intravenous thrombolysis treatment
  Interventions: Drug: alteplase
- Endovascular treatment: patient who will receive endovascular treatment
  Interventions: Procedure: endovascular

INTERVENTIONS:
Drug: acetylsalicylic acid, clopidogrel bisulfate and/or warfarin, Apixaban, Rivaroxaban, Dabigatran — subject in this group will receive oral treatment with anti platelet drug
  Other Names: Aspirin, Plavix, Coumadin, Eliquis,Xarelto, Pradaxa, Sintrom
  Groups: Conservative
Drug: alteplase — subject in this group will receive intravenous tPA
  Groups: IV tPA
Procedure: endovascular
  Other Names: subject in this group will undergo mechanical thrombectomy
  Groups: Endovascular treatment

SUMMARY:
CT perfusion (CTP) of the brain is an innovative technique to identify rapidly regions which are only partially or insufficiently perfused during an acute ischemic event. The differentiation between the core infarct and the still viable penumbra is its major clinical application. CTP helps directly in the decision-making process in the event of acute ischemic stroke by increasing the potential of success in patient who can benefit from thrombolytic/endovascular treatment.

The use of CTP in patient selection for thrombolytic/endovascular treatment was never evaluated in a prospective randomized study. Yet, clinical experience well demonstrated a good correlation between the size of the penumbra and the clinical outcome when done in early as well as late stages of the event.

The importance of identifying the penumbra in the acute phase of the ischemic stroke is widely accepted. But crucial evidence to support the predictive value of CTP to predict the clinical and anatomical/structural outcomes in the late phases (90 days after) is lacking.

Currently, the use of CTP is based on theoretical assumptions and expert opinions but a randomized prospective study to validate its use is lacking.

The current guidelines restrict the use of CTP trials and to patients that can't performed MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* NIHSS>=8
* up to 6 hours from event onset

Exclusion Criteria:

* mRS>= 3 before the start of the event
* life expectency <1 year because other disability disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women admittedto the emergency room at Rabin Medical Center, Beilinson Campus and hospitalized at the neurology department.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The predictive value of CTP in identifying penumbra (salvagable brain tissue) in event of ischemic stroke | three month

CONTACTS AND LOCATIONS:
Overall Officials: Guy Raphaeli, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tiqva, Central District, Israel

REFERENCES:
- [Background] Bivard A, Spratt N, Levi C, Parsons M. Perfusion computer tomography: imaging and clinical validation in acute ischaemic stroke. Brain. 2011 Nov;134(Pt 11):3408-16. doi: 10.1093/brain/awr257. PMID 22075524
- [Result] Koton S, Bornstein NM, Green MS. Population group differences in trends in stroke mortality in Israel. Stroke. 2001 Sep;32(9):1984-8. doi: 10.1161/hs0901.095407. PMID 11546885
- [Result] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Result] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Result] Furlan A, Higashida R, Wechsler L, Gent M, Rowley H, Kase C, Pessin M, Ahuja A, Callahan F, Clark WM, Silver F, Rivera F. Intra-arterial prourokinase for acute ischemic stroke. The PROACT II study: a randomized controlled trial. Prolyse in Acute Cerebral Thromboembolism. JAMA. 1999 Dec 1;282(21):2003-11. doi: 10.1001/jama.282.21.2003. PMID 10591382
- [Result] Wardlaw JM, Zoppo G, Yamaguchi T, Berge E. Thrombolysis for acute ischaemic stroke. Cochrane Database Syst Rev. 2003;(3):CD000213. doi: 10.1002/14651858.CD000213. PMID 12917889
- [Result] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Result] Parsons MW. Perfusion CT: is it clinically useful? Int J Stroke. 2008 Feb;3(1):41-50. doi: 10.1111/j.1747-4949.2008.00175.x. PMID 18705914
- [Result] Goyal M, Menon BK, Derdeyn CP. Perfusion imaging in acute ischemic stroke: let us improve the science before changing clinical practice. Radiology. 2013 Jan;266(1):16-21. doi: 10.1148/radiol.12112134. No abstract available. PMID 23264523
- [Result] Gonzalez RG, Copen WA, Schaefer PW, Lev MH, Pomerantz SR, Rapalino O, Chen JW, Hunter GJ, Romero JM, Buchbinder BR, Larvie M, Hirsch JA, Gupta R. The Massachusetts General Hospital acute stroke imaging algorithm: an experience and evidence based approach. J Neurointerv Surg. 2013 May;5 Suppl 1(Suppl 1):i7-12. doi: 10.1136/neurintsurg-2013-010715. Epub 2013 Mar 14. PMID 23493340
- [Result] Abstracts of the 17th European Stroke Conference. Nice, France. May 13-16, 2008. Cerebrovasc Dis. 2008;25 Suppl 2:1-204. doi: 10.1159/000132086. No abstract available. PMID 22015331